CLINICAL TRIAL: NCT05167916
Title: Can Four Weeks-check Cystoscopy and Urine Cytology After Primary Complete Resection of T1 Bladder Cancer Replace Repeat Biopsy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Lecturer of Urology, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AS-12-2021
Record Dates: First submitted 2021-11-23; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Cystoscopy; Cytology; Repeat biopsy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T1 Bladder cancer patients (Experimental)
  Interventions: Procedure: Outpatient check cytoscopy; Diagnostic Test: Urine cytology

INTERVENTIONS:
Procedure: Outpatient check cytoscopy — Four weeks after primary TURBT, study participants will provide freshly voided urine sample which will be sent for cytology assessment by uropathologist in charge according to the Paris classification system. Suspicious sample for malignancy, low- and high-grade malignant samples will be considered positive results. On the other hand, hyperplastic or negative samples for malignancy will be defined as negative results.
  Thereafter, patients will be assessed by flexible white light check cystoscopy under local anesthesia using flexible instrument by single operator. Checklist will be fulfilled by the operator urologist. Check cystoscopy will be considered positive when encountering residual gross lesion at the area of previous resection or newly developed lesions or both.
Diagnostic Test: Urine cytology — Four weeks after primary TURBT, study participants will provide freshly voided urine sample which will be sent for cytology assessment by uropathologist in charge according to the Paris classification system. Suspicious sample for malignancy, low- and high-grade malignant samples will be considered positive results. On the other hand, hyperplastic or negative samples for malignancy will be defined as negative results.
  Thereafter, patients will be assessed by flexible white light check cystoscopy under local anesthesia using flexible instrument by single operator. Checklist will be fulfilled by the operator urologist. Check cystoscopy will be considered positive when encountering residual gross lesion at the area of previous resection or newly developed lesions or both.

SUMMARY:
The primary objective of this prospective study is to evaluate the clinical performance of combined check cystoscopy and urine cytology findings 4 weeks after initial primary complete resection of T1 BC for detection of residual malignancy at repeat biopsy.

DETAILED DESCRIPTION:
Non muscle invasive bladder cancer (NMIBC) represents the vast majority (70%-80 %) of bladder cancer (BC) patients. T1 disease accounts for 15% to 30 % of NMIBC and is defined as invasion of the lamina propria without invasion of the muscularis propria.

Complete primary transurethral resection of bladder tumor (TURBT) is considered a crucial initial step not only to establish the diagnosis but also to achieve good prognosis and to guard against early recurrence due to missed lesions. Most current guidelines recommend repeat biopsy at 2 to 6 weeks after initial complete resection of T1 BC before initiation of adjuvant intravesical instillation of bacillus of Calmette and Guerin (BCG).

Repeat biopsy after presumable complete primary TURBT of T1 disease is quite helpful to confirm complete resection; in addition, it can provide additional pathological information as residual T1/Ta disease in 33%-55% of patients and T2 disease (upstaging) in 3%-10% of patients.

However, repeat biopsy is still an invasive procedure adding further cost and risk of anesthetic as well as surgical complications. In addition, it was shown in a recent published report by Adam and colleagues that repeat biopsy alters further patient management in a minority of patients and delay adjuvant intravesical BCG in 90% of patients.

Therefore, ensuring adequate primary complete resection by less invasive tools might be a helpful step to spare large proportion of T1 BC patients the added cost and morbidity of repeat biopsy, and to prioritize patients for intervention in systems with long waiting times, as well.

Urine cytology is a useful noninvasive method for detection of urothelial carcinoma of the urinary bladder. It has been established as a useful adjunct in both the diagnosis and follow-up especially for high grade tumor, and carcinoma in situ (CIS).

Urine cytology after complete primary resection of NMIBC had been investigated in previous reports as a determinant factor of possible overlooked tumors after primary resection.

On the other hand, check outpatient cystoscopy under local anesthesia remains the gold standard tool of initial diagnosis and surveillance of NMIBC. However, it lacks the sensitivity to detect flat lesions (more likely CIS).

In this context, the investigators assume that combined check outpatient cystoscopy and urine cytology 4 weeks after initial complete resection of T1 BC can provide reliable information about possibility of residual tumor/s that necessities repeat biopsy.

In the current study, the investigators aim at evaluating the clinical performance of combined check cystoscopy and urine cytology findings 4 weeks after initial primary complete resection of T1 BC for detection of residual malignancy at repeat biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged >18 years)
* Patients with primary or recurrent NMIBC for whom complete primary TURBT was done.

Exclusion Criteria:

* Patients with incomplete resection
* Patients with nonurothelial carcinoma or variant histology.
* Patient with biopsy proven muscle invasion, or Ta BC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of positive repeat biopsy for malignancy | 4 weeks
  The primary outcome include evaluation of the clinical performance of combined urine cytology and outpatient check cystoscopy 4 weeks after primary complete resection of T1BC as a predictive tool for possible residual malignancy at repeat biopsy.

SECONDARY OUTCOMES:
Tumor recurrence rate | 1 year
  The secondary outcome includes the evaluation of predictive capacity of combined urine cytology and outpatient check cystoscopy for early tumor recurrence in the study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Mansoura University
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided